CLINICAL TRIAL: NCT01227616
Title: Ferumoxytol for Anemia of CKD Trial (FACT): A Phase IV, Open-Label, Multicenter Trial, With MRI Substudy, of Repeated Doses of Ferumoxytol Compared With Iron Sucrose for Treatment of IDA in CKD Patients on Hemodialysis
Brief Title: Compare Efficacy/Safety of Repeat Doses of Ferumoxytol With Iron Sucrose in CKD Subjects With IDA and on Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMAG-FER-CKD-401
Record Dates: First submitted 2010-10-22; First posted 2010-10-25 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-03

CONDITIONS: Iron Deficiency Anemia Treatment; Chronic Kidney Disease(CKD)
Keywords: Iron deficiency anemia (IDA); chronic kidney disease (CKD); hemodialysis; magnetic resonance imaging (MRI); ferumoxytol; Feraheme
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia, Iron-Deficiency | interventions — Ferrosoferric Oxide; Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ferumoxytol (Experimental): Intravenous (IV) iron
  Interventions: Drug: Ferumoxytol
- IV Iron Sucrose (Active Comparator): Intravenous (IV) iron
  Interventions: Drug: Iron Sucrose

INTERVENTIONS:
Drug: Ferumoxytol — IV Ferumoxytol
  Other Names: Feraheme
  Arms: Ferumoxytol
Drug: Iron Sucrose — IV Iron Sucrose
  Other Names: Venofer
  Arms: IV Iron Sucrose

SUMMARY:
The objectives of this study are to compare the efficacy and safety of repeat doses of intravenous (IV) ferumoxytol with IV iron sucrose for the treatment of IDA in subjects with hemodialysis-dependent CKD.

DETAILED DESCRIPTION:
This was a Phase IV, randomized, open-label, active-controlled, multicenter clinical trial designed to evaluate the safety, efficacy, and frequency of use of ferumoxytol compared to iron sucrose for the episodic treatment of IDA in hemodialysis subjects with CKD over a 1-year period. As part of this Main Study, an Oxidative Stress Substudy and an MRI Substudy were conducted. The Oxidative Stress Substudy, to be run concurrently with the initial TP of the Main Study, was to examine the varying degrees to which iron sucrose and ferumoxytol may or may not induce oxidative stress in vitro in subjects undergoing hemodialysis. The MRI Substudy, to be run concurrently with the Main Study and continue for an additional 11 months, was to assess the potential for deposition of iron in cardiac, hepatic, and pancreatic tissues and changes in laboratory parameters over a 2-year period.

ELIGIBILITY:
Key Inclusion Criteria include:

1. Males and females ≥18 years of age
2. Diagnosis of CKD
3. Subjects on dialysis must have been on dialysis for at least 3 months prior to screening
4. Female subjects of childbearing potential who are sexually active must be on an effective method of birth control for at least 1 month prior to screening and agree to remain on birth control until completion of participation in the study

Key Exclusion Criteria include:

1. History of allergy to either oral or IV iron
2. Female subjects who are pregnant or intend to become pregnant, breastfeeding, within 3 months postpartum, or have a positive serum or urine pregnancy test
3. Parenteral iron therapy within 30 days prior to screening or red blood cell (RBC)/whole blood transfusion within 14 days prior to screening or planned during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (36):
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Pine Bluff, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Azusa, California
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Beverly Hills, California
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Lynwood, California
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Northridge, California
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Paramount, California
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Sacramento, California
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, San Gabriel, California
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Simi Valley, California
  - For additional information regarding investigative sites for this trial , contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Whittier, California
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Whittier, California
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Middlebury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Coral Springs, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Augusta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Macon, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, New Orleans, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Framingham, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Pontiac, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Roseville, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Farmington, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Brooklyn, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Ridgewood, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, The Bronx, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Asheville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Bethlehem, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Arlington, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Edinburg, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, San Antonio, Texas
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) , or speak with your personal physician, Montreal
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Montreal
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Toronto
- United Kingdom (2):
  - For additional information regarding investigative sites for this trial , contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, London
  - For additional information regarding investigative sites for this trial, contact 1-877-411-2510 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, London

REFERENCES:
- [Result] Macdougall IC, Strauss WE, Dahl NV, Bernard K, Li Z. Ferumoxytol for iron deficiency anemia in patients undergoing hemodialysis. The FACT randomized controlled trial . Clin Nephrol. 2019 Apr;91(4):237-245. doi: 10.5414/CN109512. PMID 30802204
- [Derived] Macdougall IC, Dahl NV, Bernard K, Li Z, Batycky A, Strauss WE. The Ferumoxytol for Anemia of CKD Trial (FACT)-a randomized controlled trial of repeated doses of ferumoxytol or iron sucrose in patients on hemodialysis: background and rationale. BMC Nephrol. 2017 Apr 3;18(1):117. doi: 10.1186/s12882-017-0523-8. PMID 28372549

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 296 hemodialysis patients with IDA who met the entry criteria were enrolled and randomized (ferumoxytol: n=197; iron sucrose: n=99).
  One subject in the ferumoxytol group and 2 subjects in the iron sucrose group withdrew prior to receiving study drug, resulting in 293 total participants for analysis.
Groups:
- Ferumoxytol: 30 mg Fe/mL for IV injection
- Iron Sucrose: 20 mg Fe/mL for IV injection
Period: Overall Study
Arm/Group | Ferumoxytol | Iron Sucrose
Started | 196 | 97
Completed | 142 | 74
Not Completed | 54 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ferumoxytol | Iron Sucrose | Total
Number analyzed (Participants) | 196 | 97 | 293
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (14.13) | 57.6 (13.62) | 58.8 (13.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 40 | 122
  Male | 114 | 57 | 171
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 68 | 40 | 108
  Not Hispanic or Latino | 128 | 57 | 185
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 4 | 14
  Asian | 15 | 13 | 28
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 5
  Black or African American | 62 | 26 | 88
  White | 101 | 47 | 148
  More than one race | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 185 | 90 | 275
  Canada | 5 | 2 | 7
  United Kingdom | 6 | 5 | 11
Mean Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 10.4 (0.74) | 10.4 (0.81) | 10.4 (0.76)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin Changes
Description: Changes in the mean hemoglobin between Baseline and Week 5 for ferumoxytol and iron sucrose in each treatment period.
Time Frame: Up to 6 treatment periods (5 weeks per treatment period)
Population: Mean Change in Hemoglobin at Week 5 - ITT Population
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Ferumoxytol | Iron Sucrose
Number analyzed (Participants) | 196 | 97
g/dL
  TP1: number analyzed (Participants) | 195 | 94
  TP1 | 0.5 (0.97) | 0.4 (0.97)
  TP2: number analyzed (Participants) | 167 | 88
  TP2 | 0.6 (0.96) | 0.3 (1.03)
  TP3: number analyzed (Participants) | 130 | 64
  TP3 | 0.6 (1.10) | 0.4 (0.87)
  TP4: number analyzed (Participants) | 81 | 32
  TP4 | 0.5 (1.12) | 0.6 (1.11)
  TP5: number analyzed (Participants) | 48 | 17
  TP5 | 0.4 (1.14) | 0.3 (0.96)
  TP6: number analyzed (Participants) | 22 | 8
  TP6 | 0.5 (1.21) | -0.3 (1.00)
Statistical Analysis 1: Comparison: Ferumoxytol; Test type: Non-Inferiority — The study protocol defined the margin for non-inferiority as 0.5 g/dL meaning non-inferiority would be established in a TP if the lower limit of the 95% confidence limit for the difference between ferumoxytol and iron sucrose mean change was ≥0.5 g/dL; p < 0.05, ANCOVA; Stats. of primary endpoint performed only for TP1 and TP2. 240 subjects retreated should yield 90% power to detect non-inferiority during TP2; Mean Difference (Final Values) = 0.5

2. Secondary Outcome: Changes in Transferrin Saturation (TSAT)
Description: Mean change in TSAT from TP Baseline to Week 5 for each TP
Time Frame: Up to 6 treatment periods (5 weeks per treatment period)
Population: Mean Change in TSAT at Week 5 - ITT Population
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Ferumoxytol | Iron Sucrose
Number analyzed (Participants) | 195 | 95
Percent
  TP1 | 6.6 (9.2) | 9.5 (11.97)
  TP2: number analyzed (Participants) | 169 | 88
  TP2 | 8.2 (12.95) | 11.3 (14.68)
  TP3: number analyzed (Participants) | 129 | 63
  TP3 | 8.5 (10.56) | 9.1 (11.13)
  TP4: number analyzed (Participants) | 80 | 32
  TP4 | 9.8 (14.76) | 10.0 (14.76)
  TP5: number analyzed (Participants) | 48 | 17
  TP5 | 6.3 (9.77) | 14.4 (17.05)
  TP6: number analyzed (Participants) | 21 | 8
  TP6 | 7.1 (16.62) | 5.1 (12.84)

3. Secondary Outcome: Proportion of Subjects With an Increase in Hemoglobin of ≥1.0 g/dL at Any Time From TP Baseline to Week 5 for Each TP
Description: The proportion of subjects by group achieving a ≥1.0 g/dL increase in hemoglobin at any point during each 5-week treatment period.
Time Frame: Up to 6 treatment periods (5 weeks per treatment period)
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Ferumoxytol | Iron Sucrose
Number analyzed (Participants) | 196 | 97
participants
  TP1 | 55 | 23
  TP2: number analyzed (Participants) | 173 | 88
  TP2 | 55 | 13
  TP3: number analyzed (Participants) | 133 | 65
  TP3 | 42 | 19
  TP4: number analyzed (Participants) | 85 | 33
  TP4 | 20 | 10
  TP5: number analyzed (Participants) | 49 | 18
  TP5 | 13 | 3
  TP6: number analyzed (Participants) | 22 | 8
  TP6 | 5 | 1

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events starting on or after day 0 up to 13 months
Description: Safety population included all patients who received any study drug.
Arm/Group | Ferumoxytol | Iron Sucrose
All-Cause Mortality (participants affected / at risk) | 16/196 | 6/97
Serious Adverse Events (participants affected / at risk) | 93/196 | 49/97
Other Adverse Events (participants affected / at risk) | 158/196 | 81/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferumoxytol (N=196) | Iron Sucrose (N=97)
Infections and infestations (Infections and infestations) | 38 (49) | 17 (24)
Sepsis (Infections and infestations) | 10 (10) | 2 (2)
Pneumonia (Infections and infestations) | 7 (7) | 3 (4)
Cellulitis (Infections and infestations) | 4 (4) | 2 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 25 (32) | 12 (21)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Cardiac disorders (Cardiac disorders) | 20 (31) | 15 (27)
Cardiac failure congestive (Cardiac disorders) | 5 (5) | 5 (7)
Acute myocardial infarction (Cardiac disorders) | 4 (4) | 3 (6)
Angina pectoris (Cardiac disorders) | 3 (4) | 4 (6)
Cardiac arrest (Cardiac disorders) | 3 (5) | 2 (2)
Cardio-respiratory arrest (Cardiac disorders) | 4 (4) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 18 (22) | 16 (20)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 4 (5) | 4 (4)
Hip fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 21 (27) | 6 (9)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 17 (18) | 10 (21)
Fluid overload (Metabolism and nutrition disorders) | 9 (10) | 4 (9)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (5) | 4 (6)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Vascular disorders (Vascular disorders) | 12 (14) | 13 (14)
Nervous system disorders (Nervous system disorders) | 13 (16) | 9 (12)
General disorders and administration site conditions (General disorders) | 9 (10) | 6 (6)
Non-cardiac chest pain (General disorders) | 5 (5) | 2 (2)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 7 (8) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 4 (5) | 4 (4)
Psychiatric disorders (Psychiatric disorders) | 6 (11) | 2 (3)
Mental status changes (Psychiatric disorders) | 5 (10) | 1 (2)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 3 (6) | 3 (4)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1)
Immune system disorders (Immune system disorders) | 2 (2) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Investigations (Investigations) | 0 (0) | 2 (2)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 0 (0) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ferumoxytol (N=196) | Iron Sucrose (N=97)
Gastrointestinal disorders (Gastrointestinal disorders) | 74 (163) | 36 (85)
Nausea (Gastrointestinal disorders) | 22 (30) | 15 (17)
Diarrhoea (Gastrointestinal disorders) | 21 (25) | 12 (13)
Vomiting (Gastrointestinal disorders) | 16 (20) | 12 (15)
Abdominal pain (Gastrointestinal disorders) | 12 (14) | 8 (9)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 61 (135) | 42 (101)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 14 (18) | 8 (25)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 7 (8) | 7 (7)
Fall (Injury, poisoning and procedural complications) | 7 (7) | 6 (6)
Infections and infestations (Infections and infestations) | 64 (112) | 33 (61)
Upper respiratory tract infection (Infections and infestations) | 14 (14) | 6 (7)
Urinary tract infection (Infections and infestations) | 12 (12) | 3 (3)
Pneumonia (Infections and infestations) | 11 (12) | 3 (4)
Sepsis (Infections and infestations) | 10 (10) | 2 (2)
Cellulitis (Infections and infestations) | 5 (5) | 6 (7)
General disorders and administration site conditions (Gastrointestinal disorders) | 57 (87) | 21 (37)
Non-cardiac chest pain (General disorders) | 10 (11) | 7 (12)
Pyrexia (General disorders) | 15 (17) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 40 (127) | 25 (82)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (16) | 11 (22)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 16 (70) | 7 (37)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 7 (10)
Vascular disorders (Vascular disorders) | 38 (77) | 24 (38)
Hypotension (Vascular disorders) | 17 (21) | 7 (8)
Hypertension (Vascular disorders) | 14 (37) | 6 (14)
Nervous system disorders (Nervous system disorders) | 35 (48) | 24 (48)
Dizziness (Nervous system disorders) | 10 (11) | 7 (18)
Headache (Nervous system disorders) | 8 (12) | 7 (9)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 41 (74) | 18 (30)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 5 (5)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (13) | 6 (6)
Cardiac disorders (Cardiac disorders) | 30 (64) | 18 (33)
Cardiac failure congestive (Cardiac disorders) | 6 (6) | 5 (7)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 32 (51) | 15 (29)
Fluid overload (Metabolism and nutrition disorders) | 14 (15) | 6 (12)
Hyperkalaemia (Metabolism and nutrition disorders) | 11 (11) | 5 (7)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 19 (32) | 10 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (15) | 4 (5)
Psychiatric disorders (Psychiatric disorders) | 18 (30) | 7 (11)
Investigations (Investigations) | 11 (12) | 13 (21)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 14 (20) | 6 (6)
Anaemia (Blood and lymphatic system disorders) | 8 (12) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If there is no multi-site publication within 18 months after the Study has been completed or terminated at all Study sites, and all data have been received by Sponsor, the Site, and SMO shall have the right to publish its results from the Study for non-commercial purposes, if submitted to Sponsor for review 60 days prior to submission of publication. Publication must remove all confidential information and may be delayed by up to 180 days to allow Sponsor to protect its interests.